CLINICAL TRIAL: NCT05952297
Title: A Novel Wearable Device to Improve Sleep Quality
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kelly Glazer Baron, PhD, MPH, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00165943
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Insomnia
Keywords: insomnia; sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: For the first 28 days, participants will be randomized 1:1 to intervention vs. placebo. Following 28 days, all devices will be active from day 28 to 3 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Devices will appear the same but some devices will be placebo and some will be turned on as active. This is turned on remotely. A staff member who is blinded to the study screening and outcomes will conduct the randomization allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Wellness Device (Experimental): The wearable sleep wellness device that contains specially designed coils that generate micro electromagnetic stimulation located in the neckband and is worn around the neck like headphones for at least 3 hours per day.
  Interventions: Device: Sleep Wellness Device (BeCurie)
- Inactive Sleep Wellness Device (Sham Comparator): This sleep wellness device is running an inactive program in the application (no electromagnetic stimulation).
  Interventions: Device: Sleep Wellness Device (BeCurie)

INTERVENTIONS:
Device: Sleep Wellness Device (BeCurie) — This device emits micro electromagnetic stimulation

SUMMARY:
The purpose of the study is to help determine if a wearable sleep wellness device improves sleep among adults with insomnia. This study will enroll a total of 60 participants for this remotly conducted study and randomize 1:1 for treatment and control.

Aim 1 of the study is to test the effects of the sleep wellness device compared to a placebo device on sleep after 28 days of use.

Aim 2 of the study is to test the longer term effects of the sleep wellness device at 3 month follow-up.

DETAILED DESCRIPTION:
BeCurie is a wearable sleep wellness device that contains specially designed coils that generate micro electromagnetic stimulation located in the neckband. This device is classified as a low risk wellness device that does not need FDA approval. It can be used by anyone aged 18 and above.

To test the efficacy of this device, a clinical study entitled "Prospective Observational Double-Blind Placebo-Controlled Randomised Clinical Study to Assess the Stress and Anxiety Improvement with BeCurie" was carried out. (CTRI Registration CTRI/2022/03/041445 )Compared to the placebo group, the treatment group showed improvements in all stress and anxiety-related parameters, showing the effectiveness of the BeCurie device in managing stress and anxiety in individuals with perceived stress and anxiety. Further, no changes were observed in blood profile, biochemistry, and physiological parameters in both groups. No adverse events or side effects were recorded during the study in both placebo and treatment arms, demonstrating BeCurie has been well tolerated.

Further testing is warranted to determine whether or not this device has an influence on the quality of sleep of those who wear it. Therefore the goal of this study is to test the effects of this sleep wellness device on sleep quality among adults with elevated insomnia symptoms. This study will test the sleep wellness device compared to a placebo device for changes in sleep over 28 days. Following this 28 day blinded trial, this study will study the effects of the device in an open label, one group study from 28 days to 3 months. This study is fully remote, with no in person office visits. All assessments will occur via web-based surveys, sleep wearable devices (fitbit) and text-message based sleep diaries.

ELIGIBILITY:
Inclusion Criteria:

* Clinically elevated insomnia symptoms as defined by Insomnia Severity Index (ISI) score >=15
* Able to read and write in English
* Smartphone user

Exclusion criteria:

* History of chronic drug or alcohol abuse
* More than 400mg of caffeine per day
* Consistent travel across time zones throughout the study period
* Consistent migraine attacks or headaches
* Diagnosed sleep disorders other than insomnia
* Prescribed sleep medications or other treatments for insomnia (e.g. cognitive behavioral therapy)
* Untreated or unstable psychiatric disorders as defined by a PHQ8 score of greater than 15
* Using antipsychotic drugs
* Pregnant women or lactating women, or have an infant less than 6 months old
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* A history of serious medical conditions (e.g. cancers, consistent hospitalizations)
* History of allergy or hypersensitivity to any medical device or its components
* Overnight work >1 shift per month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Anderson DJ, Troxel WM, Landvatter J, Baron KG. A randomized pilot study of a wearable device using variable complex weak magnetic fields among participants with insomnia symptoms. J Clin Sleep Med. 2025 Jul 1;21(7):1285-1291. doi: 10.5664/jcsm.11690. PMID 40165746

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sleep Wellness Device | Inactive Sleep Wellness Device
Started | 28 | 31
Completed | 27 | 31
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Wellness Device | Inactive Sleep Wellness Device | Total
Number analyzed (Participants) | 28 | 31 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (12.5) | 41.6 (11.8) | 40.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 4 | 6
  White | 20 | 22 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Symptoms
Description: The insomnia severity index (ISI) is a self-report item of insomnia symptoms that is well correlated with insomnia diagnoses, with higher scores being worse insomnia. Scores range from 0-28.
Time Frame: Change from baseline in insomnia symptoms at 28 days
Population: Data missing for 2 participants in the control group at 1 month. Data missing for 3 intervention participants at 1 month due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep Wellness Device | Inactive Sleep Wellness Device
Number analyzed (Participants) | 25 | 29
score on a scale | -7.34 (1.87) | -7.58 (.84)
Statistical Analysis 1: Comparison: Inactive Sleep Wellness Device; Test type: Superiority; p = .88, mixed model; linear mixed model, time x condition effect

ADVERSE EVENTS:
Time Frame: 3 months
Description: Participants reported adverse events to study staff
Arm/Group | Sleep Wellness Device | Inactive Sleep Wellness Device
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/31
Other Adverse Events (participants affected / at risk) | 1/28 | 3/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sleep Wellness Device (N=28) | Inactive Sleep Wellness Device (N=31)
headache (General disorders) | 1 (1) | 3 (3) — Headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT05952297/Prot_SAP_000.pdf